CLINICAL TRIAL: NCT00711191
Title: A Phase 1 Dose Escalation Open Label Study Of CP-870,893 In Combination With Gemcitabine In Patients With Chemotherapy-Naïve Surgically Incurable Pancreatic Cancer
Brief Title: A Study On An Immunostimulant Antibody In Combination With Chemotherapy For Advanced Cancer Of The Pancreas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5021005
Record Dates: First submitted 2008-06-26; First posted 2008-07-08 (Estimated); Results first posted 2012-06-06 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-11

CONDITIONS: Pancreatic Neoplasm
Keywords: pancreas cancer; cancer of the pancreas; gemcitabine; chemotherapy; monoclonal antibody; immunotherapy; CD40
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Antibodies, Monoclonal; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Experimental)
  Interventions: Biological: monoclonal antibody; Drug: chemotherapy

INTERVENTIONS:
Biological: monoclonal antibody — CP-870,893 intravenous administration [IV] on day 3 of 4-week cycles
Drug: chemotherapy — gemcitabine 1000 mg/m^2 intravenous administration [IV] q week [wk]x3 of 4-week cycles

SUMMARY:
This study aims to seek evidence that activation of certain cells of the immune system will be safe and well tolerated in combination with cytotoxic chemotherapy. Preliminary evidence of clinical anti-tumor activity will be sought.

ELIGIBILITY:
Inclusion Criteria:

* 1st-line surgically incurable cancer of the pancreas
* ECOG(Eastern Cooperative Oncology Group) performance status 0-1

Exclusion Criteria:

* Previous systemic therapy for pancreas cancer
* History of cancer-associated blood clots
* History of autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Beatty GL, Chiorean EG, Fishman MP, Saboury B, Teitelbaum UR, Sun W, Huhn RD, Song W, Li D, Sharp LL, Torigian DA, O'Dwyer PJ, Vonderheide RH. CD40 agonists alter tumor stroma and show efficacy against pancreatic carcinoma in mice and humans. Science. 2011 Mar 25;331(6024):1612-6. doi: 10.1126/science.1198443. PMID 21436454
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5021005&StudyName=A%20Study%20On%20An%20Immunostimulant%20Antibody%20In%20Combination%20With%20Chemotherapy%20For%20Advanced%20Cancer%20Of%20The%20Pancreas

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-870893 0.1 mg/kg: Participants received chemotherapy (gemcitabine) with a starting dose of 1000 milligrams per meter squared (mg/m^2) intravenously (IV) on Day 1, 8, and 15 of every 28 day cycle up to a maximum of 12 cycles. CP-870893 administered IV on Day 3 of every 28 day cycle with starting dose of 0.1 milligrams per kilogram (mg/kg) (0.1 mg/kg cohort) for up to a maximum of 12 cycles.
- CP-870893 0.2 mg/kg (Escalation Cohort): Participants received chemotherapy (gemcitabine) with a starting dose of 1000 mg/m^2 IV on Day 1, 8, and 15 of every 28 day cycle up to a maximum of 12 cycles. If 0 out of 3 or <2 out of 6 participants in the CP-870893 0.1 mg/kg cohort experienced a dose limiting toxicity in Cycle 1, subsequent participants were enrolled in the 0.2 mg/kg dose cohort and received CP-870893 0.2 mg/kg IV on Day 3 of every 28 day cycle (0.2 mg/kg escalation cohort) for up to a maximum of 12 cycles.
- CP-870893 0.2 mg/kg (MTD Expansion Cohort): Participants received chemotherapy (gemcitabine) with a starting dose of 1000 mg/m^2 IV on Day 1, 8, and 15 of every 28 day cycle up to a maximum of 12 cycles. If 0 out of 3 or <2 out of 6 participants in the CP-870893 0.2 mg/kg cohort (escalation cohort) experienced a dose limiting toxicity in Cycle 1, 0.2 mg/kg was considered the maximum tolerated dose (MTD). Additional participants were enrolled in the 0.2 mg/kg dose cohort and received CP-870893 0.2 mg/kg IV on Day 3 of every 28 day cycle (0.2 mg/kg MTD expansion cohort) for up to a maximum of 12 cycles.
Period: Overall Study
Arm/Group | CP-870893 0.1 mg/kg | CP-870893 0.2 mg/kg (Escalation Cohort) | CP-870893 0.2 mg/kg (MTD Expansion Cohort)
Started | 3 | 6 | 13
Completed | 0 | 1 | 1
Not Completed | 3 | 5 | 12
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Objective progression or relapse | 2 | 3 | 7
Not completed — Withdrawal by Subject | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-870893 0.1 mg/kg | CP-870893 0.2 mg/kg (Escalation Cohort) | CP-870893 0.2 mg/kg (MTD Expansion Cohort) | Total
Number analyzed (Participants) | 3 | 6 | 13 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (7.8) | 62.3 (13.3) | 57.4 (8.1) | 59.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 8
  Male | 2 | 3 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Any of the following during first cycle of treatment and attributable to CP-870893:
  afebrile Grade (Gr) 4 neutropenia (absolute neutrophil count [ANC] <500 cells/mm^3) ≥7 days or Gr 3 or 4 neutropenia associated with fever (1 oral temperature >38.5 degrees Celsius (C) or 3 oral temperatures >38.0 degrees C in a 24-hour period); Gr 4 thrombocytopenia or Gr 3 thrombocytopenia associated with bleeding; Gr 4 lymphopenia, if coupled with clinical consequence (such as, opportunistic infection) or any other Gr 3 hematological adverse events; ≥Gr 3 non-hematologic toxicities (except alopecia).
Time Frame: Baseline up to Cycle 1 / Day 28
Population: Safety population: all participants who received any study treatment. Cubic millimeters (mm^3).
Measure: Number; unit: participants
Arm/Group | CP-870893 0.1 mg/kg | CP-870893 0.2 mg/kg (Escalation Cohort) | CP-870893 0.2 mg/kg (MTD Expansion Cohort)
Number analyzed (Participants) | 3 | 6 | 13
participants | 0 | 0 | 1

2. Secondary Outcome: Percentage of Participants With Objective Tumor Response According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Number of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST. Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as ≥30% decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat imaging study ≥4 weeks after initial documentation of response.
Time Frame: At the end of every even-numbered cycle (cycle=28 days) up to a maximum of 12 cycles and 4 to 6 weeks following initial documentation of response
Population: Safety population; Confidence Interval (CI) calculated using exact method based on binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-870893 0.1 mg/kg | CP-870893 0.2 mg/kg (Escalation Cohort) | CP-870893 0.2 mg/kg (MTD Expansion Cohort)
Number analyzed (Participants) | 3 | 6 | 13
percentage of participants | 33.3 [0.8 to 90.6] | 16.7 [0.4 to 64.1] | 7.7 [0.2 to 36.0]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is time from baseline to death from any cause. Participants last known to be alive were censored at the date of last contact.
Time Frame: Baseline, assessed monthly until death or 7.5 months after last participant was enrolled (up to January 2011)
Population: Safety population; Kaplan-Meier estimate of time to event 95 percent confidence interval (95% CI) for 50% quartile based on Brookmeyer and Crowley Method.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- CP-870893 Combined Dose Cohorts: Participants received chemotherapy (gemcitabine) with a starting dose of 1000 mg/m^2 IV on Day 1, 8, and 15 of every 28 day cycle up to a maximum of 12 cycles. CP-870893 administered IV on Day 3 of every 28 day cycle with starting dose of 0.1 mg/kg (0.1 mg/kg cohort) for up to a maximum of 12 cycles. Subsequent participants were enrolled in the 0.2 mg/kg dose cohort and received chemotherapy on Day 1, 8, and 15 or every 28 day cycle and CP-870893 0.2 mg/kg IV on Day 3 of every 28 day cycle (0.2 mg/kg escalation cohort) for up to a maximum of 12 cycles. Additional participants were enrolled in the 0.2 mg/kg dose cohort and received chemotherapy on Day 1, 8, and 15 or every 28 day cycle and CP-870893 0.2 mg/kg IV on Day 3 of every 28 day cycle (0.2 mg/kg MTD expansion cohort) for up to a maximum of 12 cycles.
Arm/Group | CP-870893 Combined Dose Cohorts
Number analyzed (Participants) | 22
months | 8.4 [5.3 to 11.8]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is time from baseline to first progression (Prog) or death from any cause. Participants last known to be alive, had not started a new (non-protocol) cancer treatment, were Prog-free, and who had a baseline and ≥1 on-study disease assessment were censored at date of last objective disease assessment that verified lack of Prog. Participants who were off treatment prior to Prog and who had no on-study disease assessment were also censored. Prog: ≥20% increase in sum of longest dimension (LD) of target lesions from smallest sum LD recorded since treatment start or appearance of ≥1 new lesions.
Time Frame: Baseline, assessed monthly until death or 7.5 months after last participant was enrolled (up to January 2011)
Population: Safety population; Kaplan-Meier estimate of time to event 95% CI for 50% quartile based on Brookmeyer and Crowley Method. Criteria for progression also included unequivocal progression of existing nontarget lesions.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CP-870893 Combined Dose Cohorts
Number analyzed (Participants) | 22
months | 5.3 [3.6 to 7.4]

5. Secondary Outcome: Time to Progression
Description: Disease progression defined as ≥20% increase in sum LD of target lesions from smallest sum LD recorded since treatment start or appearance of ≥1 new lesions. Criteria for progression also included unequivocal progression of existing nontarget lesions.
Time Frame: Monthly until death or 7.5 months after last participant was enrolled (up to January 2011)
Population: No analyses of these parameters were performed due to the Sponsor's decision to terminate clinical evaluation of CP-870893.
Arm/Group | CP-870893 Combined Dose Cohorts
Number analyzed (Participants) | 0

6. Secondary Outcome: Maximum Serum Concentration (Cmax)
Time Frame: Cycle 1 / Day 3 pre-dose, 5 minutes after End of Infusion (EOI), and 2, 6, and 24 hours after EOI and pre-dose on Day 3 of every subsequent cycle up to a maximum of 12 cycles
Population: as for outcome 5
Arm/Group | CP-870893 0.1 mg/kg | CP-870893 0.2 mg/kg (Escalation Cohort) | CP-870893 0.2 mg/kg (MTD Expansion Cohort)
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the serum concentration time-curve from time zero to the last measured concentration. AUClast analyzed using a noncompartmental approach to estimate individual participant values.
Time Frame: Cycle 1 / Day 3 pre-dose, 5 minutes after EOI, and 2, 6, and 24 hours after EOI and pre-dose on Day 3 of every subsequent cycle up to a maximum of 12 cycles
Population: as for outcome 5
Arm/Group | CP-870893 0.1 mg/kg | CP-870893 0.2 mg/kg (Escalation Cohort) | CP-870893 0.2 mg/kg (MTD Expansion Cohort)
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change (Pre-dose to Post-dose) in Plasma Cytokine Concentrations: Pre-dose Concentration (CYTO0), Maximum Concentration (CTYOMAX)
Description: An increase in values indicates greater cytokine release from cells targeted by the antibody and may be associated with an infusion reaction. Change calculated as mean of pre-dose and maximum post-dose values.
Time Frame: Cycle 1 / Day 1 prior to gemcitabine infusion (0 hour), 5 minutes after EOI and 2, 4, 6, and 24 hours after EOI; Cycle 1 / Day 3 prior to CP-970893 infusion (0 hour), 5 minutes after EOI, and 2, 4, 6, and 24 hours after EOI
Population: as for outcome 5
Arm/Group | CP-870893 0.1 mg/kg | CP-870893 0.2 mg/kg (Escalation Cohort) | CP-870893 0.2 mg/kg (MTD Expansion Cohort)
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change (Pre-dose to Post-dose) in Plasma Cytokine Concentrations: Time of Maximum Concentration (TCYTOMAX)
Description: as for outcome 8
Time Frame: as for outcome 8
Population: as for outcome 5
Arm/Group | CP-870893 0.1 mg/kg | CP-870893 0.2 mg/kg (Escalation Cohort) | CP-870893 0.2 mg/kg (MTD Expansion Cohort)
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Total and Neutralizing Human Antihuman Antibody (HAHA) Titer
Description: HAHA assessed as an indicator of immunogenicity to CP-870893.
Time Frame: Prior to infusion of CP-870893 on Day 3 of every cycle up to a maximum of 12 cycles
Population: as for outcome 5
Arm/Group | CP-870893 0.1 mg/kg | CP-870893 0.2 mg/kg (Escalation Cohort) | CP-870893 0.2 mg/kg (MTD Expansion Cohort)
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Change (Pre-dose to Post-dose) in Bone Marrow Derived Cells (B Cell) Surface Markers: CD54, CD23, CD40, CD86, and Human Leukocyte Antigen (HLA-DR)
Description: Assess the ability of PF-870893 to activate B-cells and HLA-DR which are involved in the production of antibodies. Change calculated as mean of pre-dose and post-dose values. Positive values indicate greater presence of cells associated with antibody production.
Time Frame: Cycle 1 / Day 1 and Cycle 1 / Day 8 prior to gemcitabine infusion and 6 and 24 hours after EOI; Cycle 1 / Day 3 prior to CP-870893 infusion and 6, 24, and 48 hours after EOI
Population: as for outcome 5
Arm/Group | CP-870893 0.1 mg/kg | CP-870893 0.2 mg/kg (Escalation Cohort) | CP-870893 0.2 mg/kg (MTD Expansion Cohort)
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: 18-fluorodeoxyglucose (FDG) Positron Emission Tomography (PET) Imaging (MTD Expansion Cohort)
Description: FDG PET assessment to characterize and monitor tumors before and after study treatment; measured as a standardized uptake value (SUV). A reduction in SUV from baseline for at least 1 tumor may indicate a positive metabolic response to treatment.
Time Frame: Baseline, Week 2, Week 8, and Single Time Point (STP) PET for all PET scans after Week 8
Population: as for outcome 5
Arm/Group | CP-870893 0.2 mg/kg (MTD Expansion Cohort)
Number analyzed (Participants) | 0

13. Secondary Outcome: Carbohydrate Antigen 19-9 (CA 19-9)
Description: CA 19-9 or sialylated Lewis (a) antigen (a tumor marker). Values higher than 37 units per milliliter (U/ml) considered abnormal; higher values usually indicate greater presence of disease.
Time Frame: At the end of every even-numbered cycle (cycle=28 days) and 4 to 6 weeks following initial documentation of response
Population: as for outcome 5
Arm/Group | CP-870893 0.1 mg/kg | CP-870893 0.2 mg/kg (Escalation Cohort) | CP-870893 0.2 mg/kg (MTD Expansion Cohort)
Number analyzed (Participants) | 0 | 0 | 0

14. Other Pre Specified Outcome: Recommended Phase 2 Dose (RP2D) of CP-870893 in Participants With Advanced Pancreas Cancer
Description: Additional participants enrolled at MTD of CP-870893 to further characterize suitability for phase 2 testing. RP2D confirmed if ≤ 3 our of 12 participants in expansion cohort experience DLT in cycle 1.
Time Frame: Baseline up to time of determination of maximum tolerated dose (MTD)
Population: Safety population
Measure: Number; unit: mg/kg
Groups:
- CP-870893 Combined Dose Cohorts: Participants received chemotherapy (gemcitabine) with a starting dose of 1000 milligrams per meter squared (mg/m^2) intravenously (IV) on Day 1, 8, and 15 of every 28 day cycle up to a maximum of 12 cycles. CP-870893 administered IV on Day 3 of every 28 day cycle with starting dose of 0.1 milligrams per kilogram (mg/kg) (0.1 mg/kg cohort) for up to a maximum of 12 cycles.
  Subsequent participants were enrolled in the 0.2 mg/kg dose cohort and received chemotherapy on Day 1, 8, and 15 or every 28 day cycle and CP-870893 0.2 mg/kg IV on Day 3 of every 28 day cycle (0.2 mg/kg escalation cohort) for up to a maximum of 12 cycles.
  Additional participants were enrolled in the 0.2 mg/kg dose cohort and received chemotherapy on Day 1, 8, and 15 or every 28 day cycle and CP-870893 0.2 mg/kg IV on Day 3 of every 28 day cycle (0.2 mg/kg MTD expansion cohort) for up to a maximum of 12 cycles.
Arm/Group | CP-870893 Combined Dose Cohorts
Number analyzed (Participants) | 22
mg/kg | 0.2

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were reported from the time of the first dose of study treatment up to 28 days after last dose of study treatment.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-870893 0.1 mg/kg | CP-870893 0.2 mg/kg (Escalation Cohort) | CP-870893 0.2 mg/kg (MTD Expansion Cohort)
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/6 | 5/13
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-870893 0.1 mg/kg (N=3) | CP-870893 0.2 mg/kg (Escalation Cohort) (N=6) | CP-870893 0.2 mg/kg (MTD Expansion Cohort) (N=13)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-870893 0.1 mg/kg (N=3) | CP-870893 0.2 mg/kg (Escalation Cohort) (N=6) | CP-870893 0.2 mg/kg (MTD Expansion Cohort) (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 3
Palpitations (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 5
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 4
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 3 | 6
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 2 | 3
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 3 | 5 | 10
Vomiting (Gastrointestinal disorders) | 1 | 3 | 6
Catheter site haemorrhage (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 2
Chills (General disorders) | 1 | 0 | 5
Early satiety (General disorders) | 0 | 0 | 3
Fatigue (General disorders) | 3 | 5 | 11
Nodule (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 3 | 2 | 3
Pain (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 1 | 6
Suprapubic pain (General disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 3 | 6 | 11
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 2
Blood pressure increased (Investigations) | 1 | 0 | 1
Full blood count decreased (Investigations) | 0 | 0 | 1
Neutrophil count (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 9
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 4
Dysgeusia (Nervous system disorders) | 0 | 1 | 5
Headache (Nervous system disorders) | 0 | 0 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 1
Parosmia (Nervous system disorders) | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 2
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Endodontic procedure (Surgical and medical procedures) | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.